CLINICAL TRIAL: NCT00006132
Title: Phase III Randomized Study of Oral Acyclovir in Infants With Herpes Simplex Virus Infection Involving the Central Nervous System
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Alabama at Birmingham (Other)
Purpose: Treatment
Other Study IDs: 199/15325; UAB-CASG-103
Record Dates: First submitted 2000-08-03; First posted 2000-08-04 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Herpes Simplex
Keywords: herpes simplex virus infection; herpes virus infection; immunologic disorders and infectious disorders; rare disease; viral infection
MeSH Terms: conditions — Herpes Simplex; Herpesviridae Infections; Immune System Diseases; Communicable Diseases; Rare Diseases; Virus Diseases | interventions — Acyclovir

INTERVENTIONS:
Drug: acyclovir

SUMMARY:
OBJECTIVES: I. Determine the efficacy of long term suppressive therapy with oral acyclovir in infants with herpes simplex virus infection involving the central nervous system.

II. Determine whether neurologic outcome is improved in these patients when treated with this regimen.

III. Determine whether continuous administration of this drug suppresses recurrent skin lesions in these patients.

IV. Determine the safety of this regimen in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, placebo controlled, multicenter study. Patients are stratified according to disease (CNS disease with or without cutaneous involvement vs disseminated disease with CNS involvement).

All patients receive acyclovir IV every 8 hours on days 1-21. On day 19, patients undergo a lumbar puncture and must have a negative CSF PCR to be randomized. If patients have a positive CSF PCR on day 19, they continue to receive acyclovir IV every 8 hours. Treatment continues every 7 days with a repeat CSF PCR on the fifth day until a negative CSF PCR result is achieved. Patients are then randomized to one of two treatment arms.

Arm I: Patients receive oral acyclovir three times a day for 6 months. Arm II: Patients receive placebo. In case of cutaneous recurrence during the first 12 months of the study, patients receive open label oral acyclovir (if CSF PCR is negative) or acyclovir IV (if CSF PCR is positive) for 5 days. Patients may or may not continue on study drug following this treatment.

Patients are followed at 6, 12, 24, 36, 48, and 60 months of age.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Infants diagnosed with herpes simplex virus infection involving the central nervous system with or without evidence of viral dissemination to other organs (i.e., skin, liver, or lungs) HSV-1 or HSV-2 isolated from cutaneous lesions from any site (skin, oropharynx, cerebrospinal fluid (CSF), urine, etc.) OR Must have positive CSF polymerase chain reaction (PCR) if no cutaneous skin lesions are present and viral cultures are negative No infection limited to skin, eyes, or mouth Evidence of CNS involvement includes one or more of the following: Abnormal CSF indices for term infants (WBC greater than 22/mm3 and protein greater than 115 mg/dL) Abnormal CSF indices for preterm infants (WBC greater than 25/mm3 and protein greater than 220 mg/dL) Abnormal neuroimaging study (CT with contrast, MRI with gadolinium, or head ultrasound) Disseminated disease is defined as one or more of the following: SGPT at least 2.5 times upper limit of normal Pneumonia/pneumonitis Necrotizing enterocolitis Disseminated intravascular coagulopathy
* Birth weight at least 800 grams

--Prior/Concurrent Therapy--

* No concurrent nursing from a mother who is receiving acyclovir, valacyclovir, or famciclovir for longer than 120 hours or 5 days

--Patient Characteristics--

* Renal: Creatinine no greater than 1.5 mg/dL
* Cardiovascular: No prior grade 3 or 4 intraventricular hemorrhage
* Other: No infants known to be born to HIV positive women

Ages: 0 Years to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 132
Dates: Start 1997-06

CONTACTS AND LOCATIONS:
Overall Officials: David W. Kimberlin, Study Chair — University of Alabama at Birmingham
Locations (28):
- United States (26):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - University of Arkansas, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Children's Hospital and Health Center, San Diego, California
  - Stanford University, Stanford, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - University of Florida Health Science Center - Jacksonville, Jacksonville, Florida
  - Tulane University Medical Center, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - University of Mississippi Medical Center, Jackson, Mississippi
  - St. Louis Children's Hospital, St Louis, Missouri
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Children's Hospital, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee Medical Center at Knoxville, Knoxville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern Medical School, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - University of Manitoba-Winnipeg, Winnipeg, Manitoba